CLINICAL TRIAL: NCT00048503
Title: An Open-label, Phase 2 Study of the Farnesyl Transferase Inhibitor ZARNESTRA (R115777) as Post-consolidation Therapy for Acute Myeloid Leukemia (AML) in Patients Age 60 Years and Older.
Brief Title: Study of Tipifarnib as Postconsolidation Therapy for Acute Myeloid Leukemia in Patients 60 Years and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004033; NCT00057824 (obsolete NCT alias); NCT00723034 (obsolete NCT alias)
Record Dates: First submitted 2002-11-01; First posted 2002-11-04 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Zarnestra; Acute myeloid leukemia; Tipifarnib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tipifarnib

INTERVENTIONS:
Drug: ZARNESTRA, tipifarnib, R115777

SUMMARY:
The purpose of this study is to determine if giving tipifarnib after standard treatment will prevent leukemia from coming back (relapsing). Tipifarnib belongs to a class of drugs called Farnesyl Transferase Inhibitors (FTI). It blocks proteins that make leukemia cells grow.

DETAILED DESCRIPTION:
The study is an open-label evaluation of treatment with tipifarnib in approximately 127 subjects, 60 years and older, with AML in complete remission (CR) after consolidation therapy. Prior to enrollment, patients will receive 1 or 2 cycles of induction chemotherapy. Patients who attain a CR will receive 1 or 2 cycles of consolidation chemotherapy. Patients in postconsolidation complete remission who meet the eligibility criteria are offered enrollment in the study. Subjects enrolled in the study are treated with tipifarnib A dose-modification scheme is followed to maintain adequate specified laboratory values and to minimize other adverse events. Postconsolidation treatment with tipifarnib continues until the time of relapse, death, completion of 24 cycles of treatment, or discontinuation as advised by study doctor.

Tipifarnib, film coated, compressed tablets containing 100 mg active drug, will be administered orally at a dose of 300 mg (three 100 mg film coated tablets) taken twice a day for 21 consecutive days on a 28-day cycle schedule for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed AML
* Leukemia in remission
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Acute Promyelocytic Leukemia (APL)
* Previous History of myelodysplasia or antecedent hematologic malignancy
* Previous therapy with a farnesyl transferase inhibitor

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2002-06; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine relapse-free survival (RFS) at 1 year in patients, 60 years and older with AML, who receive tipifarnib treatment.

SECONDARY OUTCOMES:
Secondary objectives, assess: overall survival; time to relapse; the safety profile of treatment with tipifarnib; the population pharmacokinetics of tipifarnib; DNA analysis of genetic variability; RNA analysis of differential gene expression.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.